CLINICAL TRIAL: NCT06814769
Title: Hyaluronic Acid in the Management of Articular Pain
Brief Title: Hyaluronic Acid and Articular Pain
Acronym: HApain
Status: Completed | Type: Observational
Sponsor: University of Catanzaro (Other)
Responsible Party: Principal Investigator, Luca Gallelli, Clinical Professor, University of Catanzaro
Other Study IDs: HA2025
Record Dates: First submitted 2025-01-31; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cross link: cross link hyaluronic acid 1 intra-articular injection
  Interventions: Device: hyaluronic acid
- linear: linear hyaluronic acid, 3 intra-articular injections
  Interventions: Device: hyaluronic acid

INTERVENTIONS:
Device: hyaluronic acid — intra-articular administration

SUMMARY:
This is a prospective longitudinal single-center clinical study on OA patients treated with HA . Patients will be enrolled at baseline (T0) and then monitored at 90 days (T1), 180 days (T2; ), and 360 days (T3). The first efficacy end-point will be the statistically significant difference (P<0.05) in VAS scale between T2 and T0 and between T3 and T2

DETAILED DESCRIPTION:
This is a prospective longitudinal single-center clinical study on OA patients treated with HA at the Pain Medicine Room of the Clinical Pharmacology and Pharmacovigilance Operative Unit of the "Renato Dulbecco" University Hospital of Catanzaro from January 2023 to December 2024. Patients will be enrolled at baseline (T0) and then monitored at 90 days (T1), 180 days (T2), and 360 days (T3). At the beginning of the study, all enrolled patients signed the informed consent. After the enrollment (T0) and during the follow ups (T1-T3), clinical and laboratory data will be collected directly by the medical staff involved in the study and Zung SAS, Zung SDS and SF-36 questionnaires will be administered. The dedicated database evaluated and recorded any systemic or local side effects. HA will be administered at the beginning of the study (T0) in agreement with the leaflet.

The first efficacy end-point will be:

the statistically significant difference (P<0.05) in VAS scale between T2 and T0 and between T3 and T2 the statistically significant difference (P<0.05) in functional mobility and walking ability (six minutes walking test) between T2 and T0 and between T3 and T2 the statistically significant difference (P<0.05) in mood disorders (Zung SAS and Zung SDS) between T2 and T0 and between T3 and T2

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both sexes between 18 and 65 years old, with a Body Mass Index < 29 kg/m2.
2. Patients with second- or third-degree of OA
3. Patients with VAS (Visual Analogue Scale) intensities higher than 5/10 who did not respond to systemic medication therapy.
4. Patients who can comprehend the study's objectives and (adhere to the orthopedist's instructions, return for follow-up, and complete the evaluation questionnaires).
5. Patients able to provide their written informed consent to participate to the study and to use their data anonymously for scientific purposes

Exclusion Criteria:

1. presence of active malignancy of any type or history of malignancy
2. Local or systemic infection.
3. Uncooperative patient or suffering from neurological disorders, therefore unable to follow the orthopedist's instructions or unable to provide informed consent for participation in the study or who have not provided written consent.
4. Any case not described in the inclusion criteria.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: After the enrollment (T0) and during the follow ups (T1-T3), clinical and laboratory data were collected directly by the medical staff involved in the study and Zung SAS, Zung SDS questionnaires were administered. The dedicated database evaluated and recorded any systemic or local side effects, in agreement with our previous studies (Gallelli et al., 2017, 2007; Marcianò et al., 2024). HA was administered in agreement with leaflet at the beginning of the study (T0) . Before the admission to this study, all the enrolled patients received systemic treatments with NSAIDs and/or local treatment with corticosteroids, without clinical benefit. Therefore, we considered the time before the administration as control group.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
pain change | 12 months
  Numeric Pain Rating Scale: with a 0-10 points, where 0 is no pain and 10 is extreme pain
mood anxiety : zung scale | 12 months
  20-items: score 0 - 44: no anxiety; 45 - 59 moderate anxiety; 60 - 80 severe anxiety

SECONDARY OUTCOMES:
mood depression: zung scale | 12 months
  20-items: score 20 to 49: no depression; 49-59 mild; 59-69 moderate; 70 - 80 severe anxiety

CONTACTS AND LOCATIONS:
Locations (1):
- Luca Gallelli, Catanzaro, CZ, Italy